CLINICAL TRIAL: NCT05104775
Title: An Open-Label, Multi-Center, Phase I Study to Evaluate the Safety, Tolerability，Pharmacokinetic/Pharmacodynamics and Anti-tumor Activity of Tetra-specific Antibody GNC-035 in Participants With Relapsed/Refractory Hematologic Malignancy and Locally Advanced or Metastatic Solid Tumors
Brief Title: A Study of GNC-035, a Tetra-specific Antibody, in Participants With Relapsed/Refractory Hematologic Malignancy
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Sichuan Baili Pharmaceutical Co., Ltd. (Industry)
Collaborators: SystImmune Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GNC-035-101
Record Dates: First submitted 2021-10-21; First posted 2021-11-03 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Hematologic Malignancies
Keywords: Relapsed/Refractory Acute B-lymphoblastic Leukemia; Relapsed/Refractory Acute Myeloid Leukemia
MeSH Terms: conditions — Hematologic Neoplasms; Recurrence; Leukemia, Myeloid, Acute

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- study treatment (Experimental): Patients receive GNC-035 as a 24-hour continuous intravenous infusion (cIV, QD) for 2 weeks (a 2-week cycle). Participants with no intolerable AEs could continue for another three cycles.
  Interventions: Drug: GNC-035

INTERVENTIONS:
Drug: GNC-035 — Administration by intravenous infusion.

SUMMARY:
In this study, the safety, tolerability and preliminary effectiveness of GNC-035 in patients with relapsed/refractory hematologic malignancies will be investigated to assess the dose-limiting toxicity (DLT), maximum tolerated dose (MTD) or maximum administered dose (MAD) for MTD is not reached of GNC-035.

ELIGIBILITY:
Inclusion Criteria:

1. The participants could understand and sign the informed consent form, and must participate voluntarily
2. No gender limit
3. Age: ≥18 and ≤75 years old
4. Life expectancy estimated to be at least 3 months
5. Histologically or cytologically confirmed relapsed or refractory non-Hodgkin's lymphoma, relapsed/refractory chronic lymphocytic leukemia, relapsed/refractory acute B-lymphoblastic leukemia, or relapsed/refractory acute myeloid leukemia
6. For relapsed or refractory chronic lymphocytic leukemia (CLL/SLL), specifically:

   * Patients who have relapsed after at least 1 line of standard therapy or who have failed or are intolerant to standard therapy;
   * Patients with relapsed or refractory chronic lymphocytic leukemia who, in the opinion of the investigator, have none or are not suitable/intolerant to other therapies;
7. For other patients with relapsed and refractory non-Hodgkin's lymphoma. These include:

   * Patients in first relapse who still progress during second-line treatment;
   * Patients who relapsed after second-line or multi-line therapy;
   * Refractory patients are defined as those who do not respond or progress after adequate dose and full cycle of standard or current commonly selected combination therapy regimens, and do not respond or progress after replacement of second-line regimens;
   * Relapsed or refractory patients who are judged by the investigator to have no or no indication/intolerance to other therapy.
8. Relapsed or refractory acute B-lymphoblastic leukemia, including:

   * Definition of refractory ALL: failure to achieve CR after standard induction therapy for bone marrow and peripheral blood response;
   * Relapsed ALL is defined as the presence of blasts (> 5%) in the peripheral blood or bone marrow, or the presence of extramedullary disease in patients who have achieved CR; mediastinal enlargement in patients who have achieved CR.
   * Special circumstances: There is no clear classification standard for adult ALL patients with number of relapse ≥ 2, persistent extramedullary leukemia and persistent positive minimal residual disease (MRD). However, most clinical trials classified these patients as refractory cases.
   * Patients with relapsed or refractory acute B-lymphoblastic leukemia who, in the opinion of the investigator, have no or no indication/intolerance to other therapy.
9. Relapsed/refractory acute myeloid leukemia (AML), relapsed/refractory AML is defined as one of the following:

   * Initial treatment who failed to respond to 2 courses of standard regimen;
   * Patients with relapse within 12 months , consolidation and intensive treatment after complete remission;
   * Patients who relapsed after 12 months but failed to respond to conventional chemotherapy;
   * Patients with two or more recurrences;
   * Patients with persistent extramedullary leukemia;
   * Patients with relapsed or refractory acute myeloid leukemia who have no or no indication/intolerance to other therapy as judged by the investigator.
10. Patients with Philadelphia chromosome positive (Ph +) acute lymphoblastic leukemia are eligible if they are intolerant or have failed first and/or second generation tyrosine kinase inhibitors (TKIs); patients with a positive T315I mutation do not require TKI salvage
11. For non-Hodgkin lymphoma, measurable lesions on CT (any lymph node lesion ≥ 1.5 cm in long diameter or > 1.0 cm in long diameter for extranodal lesions) at screening; CLL/SLL: peripheral blood leukemia cells ≥ 5.0 × 109/L; or any lymph node lesion ≥ 1.5 cm in long diameter; WM: IgM 2 × ULN;
12. For patients with acute lymphoblastic leukemia, ≥ 5% lymphoblasts in the bone marrow by morphologic assessment
13. For patients with acute myeloid leukemia, ≥ 5% blasts in the bone marrow by morphologic assessment
14. ECOG Performance Status ≤ 2
15. Recovery from toxicities of prior anticancer therapy to ≤ Grade 1 as defined by NCI-CTCAEv5.0 (except alopecia)
16. The organ function level within 7 days before the first administration meets the following requirements:

    Bone marrow function (only for patients with non-Hodgkin's lymphoma): Neutrophils without blood transfusion, G-CSF (without long-acting whitening needles within 2 weeks) and drug correction within 7 days before screening Absolute count (ANC) ≥1.0×10^9/L (for subjects with bone marrow infiltration, ≥0.5×10^9/L); hemoglobin ≥80 g/L (for subjects with bone marrow infiltration, ≥70g /L); Platelet count ≥50×10^9/L; Liver function: In the case of no hepatoprotective drugs for correction within 7 days before screening, total bilirubin ≤ 1.5 ULN (Gilbert's syndrome ≤ 3 ULN), transaminase (AST/ALT) ≤ 2.5 ULN (tumor invasive changes in the liver) Subject ≤5.0 ULN), and/or alkaline phosphatase ≤5 ULN; Kidney function: creatinine (Cr) ≤ 1.5 ULN or creatinine clearance (Ccr) ≥ 50 mL/min (calculated by the research center); Coagulation function: fibrinogen ≥ 1.5g/L; activated partial thromboplastin time (APTT) ≤ 1.5 × ULN; prothrombin time (PT) ≤ 1.5 × ULN;
17. Female participants with fertility or male participants whose partner(s) are fertile must take effective contraceptive measures from 7 days prior to the first administration to 12 weeks after the administration. Female participants with fertility must have a negative serum/urine pregnancy test in 7 days prior to the first dose.
18. Subjects are capable and willing to comply with the visits, treatment plans, laboratory examinations and other research-related procedures stipulated in the research protocol.

Exclusion Criteria:

1. Patients who have undergone major surgery within 28 days prior to dosing in this study, or are scheduled to undergo major surgery during this study ("major surgery"is defined by the investigator)
2. Pulmonary disease ≥ grade 3 according to NCI-CTCAEv5.0: including resting dyspnea, or requiring continuous oxygen therapy; patients with current interstitial lung disease (ILD) (except for those with previous interstitial pneumonia)
3. Systemic serious infections occurred within 4 weeks before screening，including but not limited to severe pneumonia, bacteremia or serious infectious complications caused by fungi, bacteria and viruses
4. Patients with active autoimmune diseases, or patients with a history of autoimmune diseases
5. Patients complicated with other malignant tumors within 5 years before the first dose, and cured non-melanoma in situ skin cancer, superficial bladder cancer, in situ cervical cancer, gastrointestinal intramucosal cancer, breast cancer, localized prostate cancer and other cancers that are considered by the investigator to be eligible
6. Positive human immunodeficiency virus antibody (HIVAb), active tuberculosis, active hepatitis B virus infection (positive HBsAg or positive HBcAb with HBV-DNA ≥ ULN), or hepatitis C virus infection (positive HCV antibody with HCV-RNA ≥ ULN)
7. Hypertension poorly controlled on medication (systolic > 150 mmHg or diastolic > 100 mmHg)
8. Left ventricular ejection fraction ≤ 45%, or history of significant cardiac disease within 1 year
9. Patients with a history of hypersensitivity to recombinant humanized antibodies or hypersensitivity to any of the excipient components of GNC-035
10. Women who are pregnant or breastfeeding
11. Previous or concomitant central nervous system disease
12. With CNS involvement
13. Prior organ transplantation or allogeneic hematopoietic stem cell transplantation (ALLo-HSCT)
14. Autologous hematopoietic stem cell transplantation (Auto-HSCT) was performed 12 weeks before starting GNC-035 treatment
15. Are using immunosuppressive agents, including but not limited to: Cyclosporine, tacrolimus, etc. within 2 weeks before GNC-035 treatment; High-dose glucocorticoids (longer than 14 days) within 2 weeks before GNC-035 treatment , A daily stable dose of >30mg of prednisone or the same dose of other glucocorticoids);
16. Radiotherapy 4 times before starting GNC-035 treatment; chemotherapy and small molecule targeted drugs 2 weeks before treatment
17. CD19 or anti-CD22 treatment and still respond, received Amgen Belintotumomab (CD19×CD3), inotuzumab-oxazomicin (CD22-ADC) treatment within 4 weeks before treatment;
18. Received CAR-T 12 weeks prior to starting GNC-035
19. Has receivedany other clinical trial within 4 weeks prior to GNC-035 treatment
20. The investigator believes that it is not suitable to participate in other situations in this clinical trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2022-02-09 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
DLT | Up to 2 weeks
  Dose limiting toxicity
MTD or MAD | Up to 2 weeks
  Maximum tolerated dose or maximum administrated dose
TEAE | Up to 2 years
  Treatment-Emergent Adverse Event
The recommended dose for future clinical study | Up to 2 weeks
  The recommended dose for future clinical study
RP2D | Up to 2 years
  Recommended phase II dose

SECONDARY OUTCOMES:
AESI | Up to 2 years
  Adverse Events of special interest
Cmax | Up to 2 weeks
  Maximum serum concentration of GNC-035
Tmax | Up to 2 weeks
  Time to maximum serum concentration (Tmax) of GNC-035
T1/2 | Up to 2 weeks
  Half-life of GNC-035
Incidence and titer of ADA | Up to 2 years
  Anti-drug antibody
ORR | Up to 2 years
  Objective Response Rate
DCR | Up to 2 years
  Disease Control Rate
PFS | Up to 2 years
  Progression-free Survival
DOR | Up to 2 years
  Duration of Response

CONTACTS AND LOCATIONS:
Overall Officials: Weili Zhao, Principal Investigator — Ruijin Hospital
Locations (7):
- China (7):
  - Guangzhou First People's Hospital, Guangzhou, Guangdong
  - Affiliated Hospital of Guizhou Medical University, Guiyang, Guizhou
  - The Fourth Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - Union Hospital Tongji Medical College Huazhong University of Science and Technology, Wuhan, Hubei
  - Shengjing Hospital of China Medical University, Shenyang, Liaoning
  - Ruijin Hospital, Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality
  - The Second People's Hospital of Yibin, Yibin, Sichuang

IPD SHARING:
Plan to Share IPD: No